CLINICAL TRIAL: NCT01979549
Title: Adverse Events During Upper Gastrointestinal Endoscopy With and Without Sedation: a Multiple Center Report From Shanghai
Brief Title: Adverse Events During Upper Gastrointestinal Endoscopy
Acronym: AEDUGESSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pudong New Area People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, diansan su, Dr., RenJi Hospital
Other Study IDs: AEDUGESSH
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Patients Need Upper Gastrointestinal Endoscopy; Peptic Ulcer; Gastric Cancer; Esophagus Cancer; Oesophagitis
Keywords: Adverse events; Upper gastrointestinal endoscopy; Sedation
MeSH Terms: conditions — Peptic Ulcer; Stomach Neoplasms; Esophageal Neoplasms; Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sedation: patients underwent upper gastrointestinal endoscopy with sedation
- non-sedation: patients underwent upper gastrointestinal endoscopy without sedation

SUMMARY:
The primary objective is to investigate the adverse events during upper gastrointestinal endoscopy with and without sedation in Chinese population

ELIGIBILITY:
Inclusion Criteria:

* Patients will undergo upper gastrointestinal endoscopy
* Age > 18 years old
* Signed informed consent form

Exclusion Criteria:

* Pregnant
* Allergy to propofol or soybean or albumen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo the upper gastrointestinal endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Investigate the adverse events according to the Adverse event reporting tool of the world SIVA International Sedation Task Force during upper gastrointestinal endoscopy with and without sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Doctor, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (3):
- China (3):
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality